CLINICAL TRIAL: NCT00260923
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study Comparing an Eight-week Treatment of Aliskiren 75 mg, 150 mg and 300 mg to Placebo in Patients With Essential Hypertension
Brief Title: A Dose Ranging Study to Compare the Safety and Efficacy of Aliskiren in Patients With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2328
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: hypertension; aliskiren; blood pressure
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
This is a study for people diagnosed with hypertension to compare 3 doses (75 mg, 150 mg, and 300 mg) of an experimental product, aliskiren in comparison to a placebo. Each patient is in the study for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 years of age and older
* Patients who are eligible and able to participate in the study

Exclusion Criteria:

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of hypertensive encephalopathy or cerebrovascular accident.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 8 weeks
Diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Sponsor GmbH
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Puig JG, Schunkert H, Taylor AA, Boye S, Jin J, Keefe DL. Evaluation of the dose--response relationship of aliskiren, a direct renin inhibitor, in an 8-week, multicenter, randomized, double-blind, parallel-group, placebo-controlled study in adult patients with stage 1 or 2 essential hypertension. Clin Ther. 2009 Dec;31(12):2839-50. doi: 10.1016/j.clinthera.2009.12.006. PMID 20110023